CLINICAL TRIAL: NCT03148639
Title: Emotion Regulation Using Virtual Reality in Schizophrenia: a Clinical and Mechanistic Trial of Avatar Therapy for Refractory Auditory Hallucinations
Brief Title: Virtual Reality Therapy for Treatment-resistant Auditory Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Responsible Party: Principal Investigator, Alexandre Dumais, Psychiatrist, researcher, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IPPM 14-006
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Auditory Hallucination, Verbal; Treatment-resistant Schizophrenia
Keywords: auditory hallucination; schizophrenia; treatment-resistant; psychotherapy; virtual reality; avatar
MeSH Terms: conditions — Hallucinations; Schizophrenia, Treatment-Resistant; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Partial crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatar therapy (Experimental): Immediate Avatar therapy.
  Interventions: Behavioral: Avatar therapy
- Treatment-as-usual (Other): Treatment-as-usual then delayed Avatar therapy.
  Interventions: Behavioral: Avatar therapy; Other: Treatment-as-usual

INTERVENTIONS:
Behavioral: Avatar therapy — Patients will receive 6 sessions of avatar therapy consisting of 45 minute (1 session per week). The therapy will consist in prompting patients to enter in a dialogue with their persecutor to better regulate their emotional responses. Over the course of the therapy, the character of the avatar will progressively become under patients' control. More precisely, the avatar's speech and tone will gradually be changed by the therapist to echo patients' improved ability to regulate their emotions. That is, the avatar will progressively change from being abusive to becoming helpful and supportive. By doing so, the therapy will seek to reinforce patients' feeling of empowerment over their voices.
Other: Treatment-as-usual — Treatment as usual will consist of typical or atypical antipsychotic medication and regulars appointments with psychiatrists and others care team members for a period of 6 weeks.
  Arms: Treatment-as-usual

SUMMARY:
Treatment of verbal hallucinations in schizophrenia is clinically challenging for both the patient and the therapist. For the therapist, one of the main difficulties arises from the impossibility of directly communicating with the entity persecuting the patient. For the patient, the therapeutic process is challenging because it aims at getting to better cope with an entity that keeps repeating stereotyped and abusive sentences without having the emotional strength to reply to the persecutor. To help overcome these clinical challenges, virtual reality enable patients to recreate the face and the voice of their persecutor.The hypothesis is that the engagement of patients in a dialogue with an external representation of their persecutor, with the support of the therapist, would help them to gain better control over their voices.

ELIGIBILITY:
Inclusion Criteria:

* distressing auditory verbal hallucinations
* medication resistance relating to auditory verbal hallucinations (no response after 3 antipsychotics trials lasting at least 4 weeks each with a minimum of 400mg chlorpromazine equivalent)
* DSM-5 diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* any change in medication within the past 2 months;
* substance use disorder within the last 12 months
* neurological disorder or unstable and serious physical illness
* ongoing psychotic episode
* cognitive behavioural therapy for psychosis within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Psychotic Symptom Rating Scale - auditory hallucinations | Within 1 week before treatment, within 1 week after treatment, follow-up 3 months
  11-item structured interview assessing the severity of auditory hallucinations

SECONDARY OUTCOMES:
Change in Beliefs About Voices Questionnaire - Revised | Within 1 week before treatment, within 1 week after treatment, follow-up 3 months
  35-item self-report measure designed to assess key beliefs and responses people have concerning their voice
Change in Positive And Negative Syndrome Scale | Within 1 week before treatment, within 1 week after treatment, follow-up 3 months
  30-item semi-structured interview investigating overall symptoms severity of schizophrenia in the last week
Change in Beck Depression Inventory - II | Within 1 week before treatment, within 1 week after treatment, follow-up 3 months
  21-item self-report measure assessing depression symptoms over the past 2 weeks
Change in Quality of Life Enjoyment and Satisfaction Questionnaire - Short From | Within 1 week before treatment, within 1 week after treatment, follow-up 3 months
  16-item self-report scale measuring enjoyment and satisfaction experienced during the past week in various areas of daily functioning

OTHER OUTCOMES:
Change in Self-reported anxiety, fear and presence | Last 10 min of each therapy session
  3-item self-report scale, ranging from 0 (no emotion) to 10 (strongest emotion)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dumais, MD, Ph.D, Principal Investigator — Institut Philippe Pinel de Montréal
Locations (1):
- Institut Universitaire en Santé Mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No